CLINICAL TRIAL: NCT03309748
Title: Remediation of Adult Black Dental Stains by Phototherapy
Brief Title: Phototherapy Remediation of Black Stain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Chirag Sheth, Associate Professor, Cardenal Herrera University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UCHCEU INDI-1531
Record Dates: First submitted 2017-10-02; First posted 2017-10-16 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Dental Deposits; Tooth Discoloration; Dental Prophylaxis
Keywords: photodynamic therapy; black-stain; Pigmented bacteria; Tannerella forsythia
MeSH Terms: conditions — Dental Deposits; Tooth Discoloration | interventions — Dental Prophylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Dental Prophylaxis (Active Comparator): Standard dental prophylaxis
  Interventions: Procedure: Dental prophylaxis
- Dental prophylaxis + antimicrobial photodynamic therapy (Active Comparator): Dental prophylaxis + aPDT
  Interventions: Procedure: Dental prophylaxis; Device: Dental prophylaxis + antimicrobial photodynamic therapy

INTERVENTIONS:
Procedure: Dental prophylaxis — American Dental Association, Code on Dental Procedures and Nomenclature (CDT) CDT code D1110
Device: Dental prophylaxis + antimicrobial photodynamic therapy — Dental prophylaxis using American Dental Association, Code on Dental Procedures and Nomenclature (CDT) CDT code D1110 followed by two 8-minute irradiation cycles using GLO Brilliant home use whitening device (GLO ™ Science LLC, New York, USA).
  Arms: Dental prophylaxis + antimicrobial photodynamic therapy

SUMMARY:
This study investigates the remediation of black-stained tooth surfaces using antimicrobial photodynamic therapy. In this crossover trial, a cohort of patients received standard dental prophylactic cleaning to remove the black stain. Later, following the washout period, (reappearance of the black stain) received photodynamic therapy in addition to the standard cleaning. Stain-free period in each of the arms was the main outcome variable. Additional microbial plaque testing was also carried out.

DETAILED DESCRIPTION:
The standard treatment practice for black dental stain is dental prophylaxis, however this is often harmful to the enamel surface and can result in tooth sensitivity. In this study we aim to explore the application of antimicrobial photodynamic therapy (aPDT) for the treatment of adult black dental stain. aPDT has demonstrated positive results in the treatment of periodontitis.

Patients received an oral examination and the extent of black stain was scored (score 1, pigmented spots or incomplete lines parallel to the gingival margin, score 2: solid lines pigmented, readily observable and limited to the cervical third of the tooth surface, score 3: pigmentation extending beyond the cervical third). The patients' oral cavity was photographed in sextants, along with a complete picture of the jaw (lingual plane) and the maxillary arch (palatal plane). For bacterial analysis, 1mg of black plaque was collected by scraping with a plastic scaler from buccal tooth surfaces taking care to avoid unnecessary removal of enamel hydroxyapatite. The first dental prophylaxis was performed to remove the black stain.

Patients were reviewed monthly and in each visit, were photographed as previously described, and the level of pigmentation scored according to the mentioned criteria. The monthly visits were continued until the black stain score returned to the initial value. The period between the first and the last appointment was noted. At this point, each volunteer received dental prophylaxis once again, followed by the application of aPDT. Antimicrobial photodynamic therapy was applied to 31 orally healthy volunteers with black stained teeth, using the GLO home whitening device (GLO™ Science LLC, New York, USA) in 2 cycles of 8 minutes. Outcome variables were area, color and time taken to reappearance of black stain following dental prophylaxis with and without antimicrobial photodynamic therapy. Differences in bacterial composition of black stain (specifically Aggregatibacter actinomycetemcomitans, Tannerella forsythia and Porphyromonas gingivalis) were analyzed DNA extracted from plaque samples. Following the application of aPDT, patients were reviewed monthly until the black stain score returned to the initial value.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with black stained (plaque on) teeth

Exclusion Criteria:

* Children
* Pregnant women
* Volunteers having completed antibiotic therapy during 15 days prior to the start of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-05-05 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
Restoration period | The period of time required for the restoration of the black stain to pre-cleaning levels will be determined by measurements carried out during Weeks 18-24, post-application of each treatment arm
  Time to restoration of the black stain following each treatment arm

SECONDARY OUTCOMES:
Black stain color | The depth of color of the black stain will be measured at Week 20 following the application of each treatment arm
  Color of the black stain
Black stain area | Area covered by the black stain will be carried out at Week 20 following the application of each treatment arm
  Area covered by the black stain
Microbial composition | Black plaque sampling will be carried out at Week 0, followed by a second sampling at Week 20, following the application of each treatment arm, in accordance with the reappearance rate of the black stain in each study volunteer
  Microbial composition of the black plaque

CONTACTS AND LOCATIONS:
Overall Officials: Maria del Mar Jovani Sancho, PhD, Study Director — Cardenal Herrera University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Albelda-Bernardo MA, Jovani-Sancho MDM, Veses V, Sheth CC. Remediation of adult black dental stains by phototherapy. BDJ Open. 2018 Apr 11;4:17035. doi: 10.1038/s41405-018-0001-9. eCollection 2018. PMID 29977603